CLINICAL TRIAL: NCT00398411
Title: Double-blind, Randomized, Mono-center, Placebo-controlled Pilot Study to Investigate the Efficacy and Safety of Moxifloxacin in the Prevention of Bacteremia After High-dose Chemotherapy and Transplantation of Peripheral Stem Cells
Brief Title: Moxifloxacin in the Prevention of Bacteremia After High-dose Chemotherapy and Transplantation of Peripheral Stem Cells
Acronym: MoxiProph
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Oliver Cornely, MD, Medical Director of the Center of Clinical Trials (ZKS), University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 05001; 2005-003271-21 (EudraCT Number)
Record Dates: First submitted 2006-11-08; First posted 2006-11-10 (Estimated); Results first posted 2013-12-11 (Estimated); Last update posted 2015-06-29 (Estimated); Status verified 2015-06

CONDITIONS: Hodgkin Disease; Non-Hodgkin Lymphoma; Multiple Myeloma; Bacteremia
Keywords: prophylaxis; bacteremia; moxifloxacin; stem cell transplantation; Hodgkin disease; non-Hodgkin lymphoma; multiple myeloma; solid tumor; autologous stem cell transplantation
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, Non-Hodgkin; Multiple Myeloma; Bacteremia | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moxifloxacin (Experimental): moxifloxacin 400 mg tablets once daily
  Interventions: Drug: moxifloxacin
- Placebo (Placebo Comparator): identical appearing placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: moxifloxacin — 400 mg p.o. per day
  Other Names: Avalox
  Arms: Moxifloxacin
Drug: placebo — one tablet per day p.o.
  Other Names: placebo preparation
  Arms: Placebo

SUMMARY:
This study investigates whether the prophylactic use of moxifloxacin during high-dose chemotherapy followed by autologous stem cell transplantation reduces the incidence of clinically significant bacteremia.

Further investigations include time to occurrence of fever, duration of fever, overall survival and antibiotic sensitivity of blood isolates.

DETAILED DESCRIPTION:
Because fluoroquinolones have broad antimicrobial coverage, bactericidal activity, high tissue concentrations, oral bioavailability and adequate tolerability and safety profiles, they are ideal candidates as antibacterial prophylaxis in cancer patients. Randomized trials investigating the effect of an antibiotic prophylaxis on patients with intermediate neutropenia have recently been conducted with levofloxacin. The influence of moxifloxacin on the incidence of bacteremia in patients undergoing autologous hematopoetic stem cell transplantation has not been investigated. Moxifloxacin may be another promising alternative, covering a broader spectrum of gram-positive and anaerobic bacteria than first- or secondary generation fluoroquinolones and for instance it is an agent administered only once daily, thus optimizing compliance, a crucial issue in prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* High-dose chemotherapy followed by peripheral autologous stem cell transplantation
* Underlying disease: Hodgkin Disease, non-Hodgkin-lymphoma, multiple myeloma or solid tumor

Exclusion Criteria:

* Allogenic stem cell transplantation
* Aplastic anemia
* Antibiotic treatment within seven days prior to randomization
* Signs and symptoms of current infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2006-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oliver A. Cornely, MD, Principal Investigator — Universität zu Köln
Locations (1):
- Klinikum der Universität zu Köln, Cologne, Germany

REFERENCES:
- [Result] Vehreschild JJ, Moritz G, Vehreschild MJ, Arenz D, Mahne M, Bredenfeld H, Chemnitz J, Klein F, Cremer B, Boll B, Kaul I, Wassmer G, Hallek M, Scheid C, Cornely OA. Efficacy and safety of moxifloxacin as antibacterial prophylaxis for patients receiving autologous haematopoietic stem cell transplantation: a randomised trial. Int J Antimicrob Agents. 2012 Feb;39(2):130-4. doi: 10.1016/j.ijantimicag.2011.10.009. Epub 2011 Dec 12. PMID 22169408

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient in: Oct 10, 2006; Last patient, last visit: Dec 08, 2008
Pre-assignment Details: 68 patients were intended for inclusion in the trial. Two patients were excluded due to violation of inclusion/exclusion criteria; both received no study drug and they were excluded from the analysis. The remaining 66 participants were evaluable for response analysis in the intention to treat (ITT) set.
Period: Overall Study
Arm/Group | Moxifloxacin | Placebo
Started | 34 | 32
Completed | 34 | 31
Not Completed | 0 | 1
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Moxifloxacin | Placebo | Total
Number analyzed (Participants) | 34 | 32 | 66
Age, Continuous [Median (Full Range); unit: years] | 54 [21 to 68] | 50 [23 to 70] | 51.5 [21 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 25
  Male | 20 | 21 | 41
Height [Mean (Standard Deviation); unit: cm] | 172.71 (8.7) | 173.72 (9.7) | 173.2 (9.1)
Weight [Mean (Standard Deviation); unit: kg] | 76.41 (13.9) | 75.00 (16.5) | 75.73 (15.1)
Underlying Disease [Number; unit: participants]
  Hodgkin's Disease | 4 | 5 | 9
  NHL | 14 | 14 | 28
  Multiple Myeloma | 16 | 12 | 28
  Solid Tumor | 0 | 1 | 1
Status of Underlying Disease [Number; unit: participants]
  primary | 20 | 14 | 34
  primary progressive | 3 | 3 | 6
  relapsed | 11 | 15 | 26

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Clinically Significant Bacteremia
Description: Failure was defined as clinically significant bacteraemia occurring in the period of neutropenia and an intervention with a systemic antibacterial becoming necessary.
  With this being a discontinuation criteria and the outcome being measured at end of treatment, only one episode is taken into account for each participant.
Time Frame: end of treatment (mean duration of treatment was 9.7 days; 10.2 days in moxifloxacin arm, 9.2 days in placebo arm)
Population: intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Moxifloxacin | Placebo
Number analyzed (Participants) | 34 | 32
participants | 3 | 9

2. Secondary Outcome: Type of Isolates and Infections
Time Frame: end of treatment (mean duration of treatment was 9.7 days; 10.2 days in moxifloxacin arm, 9.2 days in placebo arm)
Population: intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Moxifloxacin | Placebo
Number analyzed (Participants) | 34 | 32
participants
  bacteremia isolate: enterococcus faecalis | 0 | 2
  bacteremia isolate: escherichia coli | 1 | 3
  bacteremia isolate: klebsiella pneumoniae | 0 | 1
  bacteremia isolate: pseudomonas aeruginosa | 1 | 0
  bacteremia isolate: staphylococcus aureus | 1 | 1
  bacteremia isolate: staphylococcus epidermidis | 0 | 1
  bacteremia isolate: streptococcus species | 0 | 1
  clostridium difficile infection | 1 | 1
  mucositis | 0 | 1

3. Secondary Outcome: Time to Occurrence of Fever >= 38°C
Time Frame: end of treatment (mean duration of treatment was 9.7 days; 10.2 days in moxifloxacin arm, 9.2 days in placebo arm)
Population: intention to treat (ITT)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Moxifloxacin | Placebo
Number analyzed (Participants) | 34 | 32
days | 9.50 (4.1) | 7.69 (3.1)

4. Secondary Outcome: Reason for Discontinuation of Treatment
Description: Absolute neutrophil count (ANC) recovered to > 500 /µl on two consecutive days Maximum of 20 days of treatment Occurrence of fever >= 38°C Systemic antibiotic treatment despite patient being afebrile Death Other adverse event (AE) Other reason
Time Frame: end of treatment (mean duration of treatment was 9.7 days; 10.2 days in moxifloxacin arm, 9.2 days in placebo arm)
Population: intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Moxifloxacin | Placebo
Number analyzed (Participants) | 34 | 32
participants
  recovery of absolute neutrophil count | 6 | 0
  maximum of 20 days of treatment | 0 | 0
  premature discontinuation: occurence of fever | 18 | 23
  premature discontinuation: antibiotic treatment | 1 | 1
  premature discontinuation: death | 0 | 1
  premature discontinuation: other adverse event | 6 | 2
  premature discontinuation: other reason | 3 | 5

5. Secondary Outcome: Type of Infection
Time Frame: follow up visit (at discharge from hospital up to a maximum of 28 days after transplantation)
Population: intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Moxifloxacin | Placebo
Number analyzed (Participants) | 34 | 32
participants
  peri-anal abscess | 0 | 1
  mucositis | 1 | 1
  pulmonary infiltrate | 1 | 0
  infection at venous catheter | 1 | 1
  herpes infection | 8 | 8
  candida infection | 1 | 0
  acute respiratory syndrome | 1 | 0
  clostridium difficile infection | 0 | 1
  atypical pneumonia | 0 | 1

6. Secondary Outcome: Overall Survival
Time Frame: follow up visit (at discharge from hospital up to a maximum of 28 days after transplantation)
Population: intention to treat (ITT)
Measure: Number; unit: participants
Arm/Group | Moxifloxacin | Placebo
Number analyzed (Participants) | 34 | 32
participants | 34 | 31

ADVERSE EVENTS:
Time Frame: Adverse events (AE) have been documented throughout study duration, serious adverse events (SAE) until 4 weeks after end of study.
Description: The following AE have been documented in the trial but are not reported in this section unless as SAE:
  Infections, already reported as outcome measures.
  Expected AE as defined in the protocol: leukopenia, anemia, thrombocytopenia, including their manifestations; hepatosplenomegaly, bone pain, increase of lactate dehydrogenase, hyperuricemia.
Arm/Group | Moxifloxacin | Placebo
Serious Adverse Events (participants affected / at risk) | 2/34 | 3/32
Other Adverse Events (participants affected / at risk) | 34/34 | 32/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moxifloxacin (N=34) | Placebo (N=32)
atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
staphyloccocus epidermidis sepsis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Moxifloxacin (N=34) | Placebo (N=32)
abdominal cramps (General disorders) | 2 (2) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
constipation (Gastrointestinal disorders) | 8 (8) | 7 (7)
cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6)
cramps in the calf (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
diarrhea (Gastrointestinal disorders) | 26 (36) | 21 (23)
dysuria (Renal and urinary disorders) | 2 (2) | 3 (3)
edema (General disorders) | 26 (37) | 26 (42)
exanthema (Skin and subcutaneous tissue disorders) | 7 (7) | 6 (6)
fever (Infections and infestations) | 27 (35) | 31 (45)
headache (General disorders) | 10 (13) | 10 (11)
heartburn / reflux (Gastrointestinal disorders) | 6 (6) | 2 (2)
hypertension (Vascular disorders) | 2 (2) | 3 (4)
hypokalemia (General disorders) | 25 (35) | 22 (28)
hyponatremia (General disorders) | 3 (3) | 2 (2)
hypotension (Vascular disorders) | 3 (3) | 7 (7)
increase of CRP (Blood and lymphatic system disorders) | 8 (8) | 4 (4)
increase of bilirubin (Hepatobiliary disorders) | 3 (4) | 2 (4)
increase of creatinine (Renal and urinary disorders) | 0 (0) | 2 (2)
increase of liver enzymes (Hepatobiliary disorders) | 10 (20) | 13 (25)
nausea (Gastrointestinal disorders) | 31 (52) | 24 (42)
pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
vomiting (Gastrointestinal disorders) | 24 (32) | 20 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes